CLINICAL TRIAL: NCT05097677
Title: ORCHESTRA WP2 - Follow-up of Covid-19 Long Term Sequelae
Brief Title: Follow-up of Covid-19 Long Term Sequelae
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: University of Bologna (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Universiteit Antwerpen (Other); University of Sao Paulo (Other); Barcelona Institute for Global Health (Other); Fondation pour la Recherche Médicale (Other); Andaluz Health Service (Other Government); Charite University, Berlin, Germany (Other); CINECA consorzio universitario italiano (Unknown); University Medical Center Groningen (Other); Hospital Universitario Virgen Macarena (Other)
Responsible Party: Principal Investigator, Evelina Tacconelli, Professor, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: ORCHESTRA WP2
Record Dates: First submitted 2021-08-16; First posted 2021-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Acute Bronchitis; COVID-19 Acute Respiratory Distress Syndrome; COVID-19 Lower Respiratory Infection; Covid19; Corona Virus Infection; Coronavirus; Coronavirus Infections; SARS-CoV2 Infection; SARS-CoV-2 Acute Respiratory Disease; SARS-Associated Coronavirus; SARS Pneumonia; SARS (Severe Acute Respiratory Syndrome); SARS (Disease); Coronavirus Pneumonia; Coronavirus Disease 2019; Coronavirus Sars-Associated
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome; Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — COVID-19 biological samples (including blood, naso-pharingeal swabs, urine, and stool) will be collected and stored in the biobank of each participating center according to local authority regulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable (observational study) — Not applicable (observational study)

SUMMARY:
The protocol, in accordance with the objectives of ORCHESTRA project - Work Package 2, aims at investigating the characteristics and determinants of COVID-19 long-term sequelae. This goal will be reached through the harmonization of follow-up strategies across the participating cohorts to allow a standardized collection of data on COVID-19 long-term sequelae. The result will be a platform including a set of data and biomaterials from large scale international cohorts, that will be uniformly recorded, prospectively tracked and analysed. The ultimate goal will be that of providing evidence to contribute to the optimization and improvement of the management and prevention of COVID-19 sequelae.

The follow-up will be organized in multiple levels of tests, according to the capability of each cohort, and will include questionnaires to collect demographic, epidemiological and clinical data, physical examination, radiological exams and biological sampling. The long-term follow-up will also allow the assessment of long-term immunological response to SARS-CoV-2 infection and its association to the vaccination and to different treatment strategies, including monoclonal antibodies.

DETAILED DESCRIPTION:
Study design

This is a multicenter, observational, concurrent cohort study investigating COVID-19 sequelae in hospitalised and non-hospitalised patients up to 18 months after the diagnosis of SARS-CoV-2 infection.

Patients will be recruited in multiple European and non-European countries, accounting for the participation of approximately 7500 individuals in the prospective follow-up data collection.

Collection of clinical data, administration of questionnaires, collection of biological samples and imaging will take place at fixed time-points to allow a comprehensive follow-up of COVID-19 patients. The follow-up will include two levels of assessments: the first one is mandatory, the second one will be customized according to the feasibility of each cohort. An ad hoc database will be provided to each COVID-19 cohort involved to allow homogeneous and standardized data collection.

ORCHESTRA has received funding from the European Union's Horizon 2020 research and innovation programme under grant agreement No 101016167.

The Main objectives of the study are:

* To describe characteristics of COVID-19 sequelae, including type, rate, and length, through clinical, laboratory, and radiological assessments;
* To investigate valuable, confounder-adjusted, associations between COVID-19 sequelae and COVID-19 severity, comorbidities, aetiology (SARS-CoV-2 variants), treatment (including monoclonal antibodies), and trends in SARS-CoV-2 antibodies;
* To describe the rate, the aetiology (SARS-CoV-2 variants), severity, and clinical determinants of COVID-19 re-infections.

Furthermore, data retrieved from COVID-19 cohorts will allow the following:

* To compare the time course of the immunological response of the population with sequelae with the immunological response of the population without sequelae;
* To investigate immunological patterns related to specific long-term sequelae;
* To investigate possible associations of SARS-CoV-2 variants with COVID-19 severity, time course of the immunological response, and long-term sequelae;
* To describe the rate and severity of sequelae and immunological trends of COVID-19 in patients vaccinated against SARS-CoV-2;
* To describe the time course of intestinal and pulmonary microbiome after SARS-CoV-2 infection;
* To investigate possible associations of long-term sequelae with hypercoagulability;
* To describe the relationship between risk perception of reinfection and the adherence to preventative measures over time after the SARS-CoV-2 infection, including vaccine acceptance;
* To describe the use of health care services among patients recovered from SARS-CoV-2;
* To identify human and viral genetic markers indicative of disease severity using WGS or WES followed by functional analysis of the most promising variants.

Recruitment strategy

Inpatients will be recruited by the study team at the treating hospital. Outpatients will be recruited by the study team in the emergency rooms, outpatient clinics, and through the coordination with regional primary care networks.

Patients will be followed up for up to 18 months after the SARS-CoV-2 infection diagnosis. The recruitment can take place at any time between the SARS-CoV-2 infection diagnosis and the end of the 18-month follow-up, provided that the patient ensures at least one follow-up visit. Discharged inpatients as well as recovered outpatients will be invited to participate by a phone call (which will be repeated once in case of no reply). The screening/baseline data collection (including the informed consent process) can be carried out on the same day of a follow-up visit.

Before the first patient is recruited at a location, the responsible investigator will ensure that all legal and regulatory requirements are met. Patients can revoke their consent to participate in the study without restriction at any time and at their own request, without giving reasons and without any consequences for their future treatment.

Patients will be recruited by the cohort of University of Verona (UNIVR), the cohort of University of Bologna (UNIBO), the French Covid-19 cohort (INSERM), COVID-HOME study from University Medical Center Groningen (UMCG), Fondation Congolaise pour la Recherche Médicale (FCRM) cohort - Republic of The Congo, Servicio Andaluz de Salud (SAS) cohort, the cohort of the Hospital Universitario Virgen Macarena (HUVM), the cohort of Universidade Federal de São Paulo (UNIFESP)

Study procedures

This study aims to improve the COVID-19 patient care in the context of routine clinical care. Considering the lack of standardized follow-up pathways for COVID-19 patients, the selection of assessments has been based on available evidence and according to the definition of good clinical practice.

The organization of follow-up visits will be up to each center, according to the facilities and logistics of outpatient monitoring.

The follow-up will last 18 months. Day 0 corresponds to the time of the first positive SARS-CoV-2 test. The screening/baseline data collection (including the informed consent process,) can be carried out on the same day of a follow-up visit. Procedures conducted as part of the participant's routine clinical management at the time of SARS-CoV-2 active infection and obtained before the signature of the informed consent form may be recorded, provided that the procedures meet the criteria specified in the protocol.

Follow-up visits will occur at the following time-points: 3, 6, 12, 18 months. During each time-point, epidemiological data collection (SARS-CoV-2 vaccination status), treatment data collection (comorbidity management), clinical assessments (relevant medical new events, COVID-19 symptom assessment, physical examination, vital signs, 6-minute walking test), and the administration of questionnaires on functional status, respiratory impairment, and mental health will be performed as part of level I (mandatory) assessments, as well as the assessment of the SARS-CoV-2 immunological status (SARS-CoV-2 antibodies). A SARS-CoV-2 molecular test will be repeated only if positive at the previous follow-up visit. Self-administered questionnaires on symptoms, will be completed daily by the participant to provide timely data on the symptom length.

Level II (imaging, biochemistry, pulmonary function tests, electrocardiography) will be performed according to the capability of each cohort and will be based on the clinical evaluation, according to the participant's healthcare status. Imaging and biochemistry tests will be reassessed only if outside the normal ranges at the previous follow-up visit or if clinically indicated.

COVID-19 biological samples (including blood, naso-pharingeal swabs, urine, and stool) will be collected and stored in the biobank of each participating center (according to local ethic commission recommendations). Test to be performed in a centralised laboratory (genomic, transcriptomic, cytokine, viral analyses, PBMCs and genetic and epigenetic) will be sent, following international regulation, to the University of Antwerp, INSERM, University of Bologna or HMGU. Stool sample for microbiological analysis will be sent to the University of Bologna. Whole blood samples for epigenetic and genetic analysis will be sent out to UNIBO, INSERM and Helmholtz Zentrum Munchen (HMGU). In-depth human genetic analysis will be conducted using WGS or whole exome sequencing (WES) followed by functional analyses of the most promising variants. Genome-wide methylation analyses of COVID-19-positive patients in addition to a small number of control patients will enable differentiation of inherited and acquired genomic regulatory features through COVID-19 infection, which result in severe disease or an efficient clearing of infection through immune responses.

Sample size calculation

The number of inclusions will depend on the progress of the SARS-CoV-2 pandemic, which is unknown, at this time. Therefore, the number of patients who will be included cannot be determined in advance. However, depending on the timing of the project and the included cohorts, the expected enrollment is around 10000 subjects.

Statistical analysis

A comprehensive descriptive analyses taking into account sociodemographic factors and clinical courses will be carried out. The frequency distributions of the characteristics will be given in absolute and relative numbers, median plus interquartile range (IQR) or mean values plus 95% confidence interval (CIs). Associations with specific treatment strategies, disease severity patterns and laboratory results will be analysed using chi-square tests, t-tests or Mann-Whitney tests, depending on the data. To evaluate potential risk factors, multivariate regression models will be carried out. Outcome time analyses using Cox proportional-hazards regression models with time-dependent covariates will be performed to examine factors associated with each endpoint (including death). In addition, cumulative incidence functions, such as the Fine-Gray subdistribution hazard regression model, will be used to account for competing events (i.e., relocation, discharge against medical advice, etc.). For missing values, a different strategy to understand the causes and the significance for the analysis will be developed and a graduated procedure for dealing with censorship and imputations via linked regressions will be developed. The significance level is defined with a p-value <0.05. All statistical analyses will be carried out with STATA, Python and/or R statistics software by trained staff (epidemiologists, statisticians) using the latest analysis methods.

Data collection

Patient data will be collected through a specific eCRF created for the study, which will not contain personal data suitable for identifying the patient. The clinical and outcome information collected in relation to the study will be limited to the objectives of the study, taking care to reduce as much as possible the burden for the patient and for the enrolling clinical center. Only the enrolling clinical center will have access to the patient's identity and will be able to contact him if the coordinating center needs to have further information or for follow-up appointments during or after the closure of the study. For each patient, a special unique digital identification code (barcode) will be provided. The code will consist of a three-character part to identify the recruiting center and a second part consisting of 5 digits to identify the enlisted person. The code will be associated with the patient by the clinical center, which will keep a copy of it in the patient file and in the medical record. Each patient enrolled will have a specific study file with all ethical and clinical documentation. The manual for compiling the eCRF will be provided in the Trial Master File.

The data will be entered directly into the patients' eCRF and the related clinical and outcome information will be digitized in a specific database that will be developed using the RedCap® data capturing platform.

Data quality assurance

All participant data related to the study will be recorded on printed or eCRF, unless transmitted to the Sponsor or designed electronically (eg, laboratory data). The Investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the eCRF or paper CRF. The Investigator must maintain accurate documentation (source data) that supports the information entered in the eCRF or paper CRF.

The Investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents. The Promotor is responsible for the data management of this study including quality checking of the data. All source documents must be accurate, clear, unambiguous, permanent, and capable of being audited. All source documents should be made using some permanent form of recording (typing, printing, optical disc). All source documents should not be obscured by correction fluid or have temporary attachments (such as removable self-stick notes). Source documents are original records in which raw data are first recorded. These may include hospital/clinic/general practitioner records, charts, diaries, x-rays, laboratory results, pharmacy records, care records, ECG or other printouts, questionnaires, or video, for example. Source documents should be kept in a secure, limited access area.

ELIGIBILITY:
Inclusion Criteria:

* Any comorbidity
* Laboratory confirmed SARS-CoV-2 infection by PCR diagnosis from nasopharynx, oropharynx, bronchoalveolar lavage, stool, or blood. Rapid tests are an acceptable alternative.
* Individuals (or attorney or deputy who has been authorized to make the decision for patients who lack capacity) consent to participate
* Individuals over 14 years of ages

Exclusion Criteria:

* Lack of consent to participate
* Lack of laboratory confirmed SARS-CoV-2 infection.
* Individuals under 14 years of ages

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with any comorbidity with previous diagnosis of SARS-CoV-2 infection admitted to or treated as inpatients or outpatients in university and non-university hospitals or medical practices.
Sampling Method: Probability Sample
Enrollment: 7599 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical assessments of COVID-19 sequelae | 18 months
  Type of COVID-19 sequelae
Laboratory assessments of COVID-19 sequelae | 18 months
  laboratory values out of the normal ranges identified by each local laboratory
Radiological assessments of COVID-19 sequelae | 18 months
  Radiological exams described as abnormal with new findings
Length of COVID-19 sequelae | 18 months
  Days of persistence of COVID-19 sequelae
Association between SARS-CoV-2 variants and COVID-19 sequelae | 18 months
  SARS-CoV-2 variants
Association between immunological patterns and COVID-19 sequelae | 18 months
  Serological assays for virus specific neutralizing and non-neutralizing antibodies
COVID-19 reinfections | 18 months
  Rate of COVID-19 reinfections
Patterns of intestinal microbiome after SARS-CoV-2 infection | 18 months
  Metagenomic sequencing on rectal swabs/stools
Patterns of pulmonary microbiome after SARS-CoV-2 infection | 18 months
  Metagenomic sequencing on NP swabs
Human and viral genetic markers related to disease severity | 18 months
  Whole-genome sequencing or whole-exome sequencing followed by functional analysis of the most promising variants.

CONTACTS AND LOCATIONS:
Overall Officials: Evelina Tacconelli, Professor, Study Director — Universita di Verona
Locations (7):
- University of Antwerp - Laboratory of Medical Microbiology, Antwerp, Belgium
- INSERM, Paris, France
- Italy (2):
  - Policlinico S.Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- UMCG, University of Groningen, Groningen, Netherland, Netherlands
- Fondation Congolaise pour la Recherche Médicale, Brazzaville, Republic of the Congo
- Hosp. Univ. Virgen Macarena / Universidad de Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gentilotti E, Gorska A, Tami A, Gusinow R, Mirandola M, Rodriguez Bano J, Palacios Baena ZR, Rossi E, Hasenauer J, Lopes-Rafegas I, Righi E, Caroccia N, Cataudella S, Pasquini Z, Osmo T, Del Piccolo L, Savoldi A, Kumar-Singh S, Mazzaferri F, Caponcello MG, de Boer G, Hara GL; ORCHESTRA Study Group; De Nardo P, Malhotra S, Canziani LM, Ghosn J, Florence AM, Lafhej N, van der Gun BTF, Giannella M, Laouenan C, Tacconelli E. Clinical phenotypes and quality of life to define post-COVID-19 syndrome: a cluster analysis of the multinational, prospective ORCHESTRA cohort. EClinicalMedicine. 2023 Jul 21;62:102107. doi: 10.1016/j.eclinm.2023.102107. eCollection 2023 Aug. PMID 37654668

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT05097677/Prot_SAP_000.pdf